CLINICAL TRIAL: NCT02335983
Title: Phase 1b Study of Carfilzomib Administered Once Weekly in Combination With Lenalidomide and Dexamethasone in Subjects With Multiple Myeloma
Brief Title: Phase 1b Study of Weekly Carfilzomib in Combination With Lenalidomide and Dexamethasone in Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFZ013
Record Dates: First submitted 2014-12-23; First posted 2015-01-12 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; WW Domain-Containing Oxidoreductase; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- RRMM Dose-evaluation: Carfilzomib 56 mg/m² (Experimental): Participants with relapsed or refractory multiple myeloma (RRMM) received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 56 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- RRMM Dose-evaluation: Carfilzomib 70 mg/m² (Experimental): Participants with RRMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- RRMM Dose-expansion: Carfilzomib 70 mg/m² (Experimental): Participants with RRMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² (Experimental): Participants with newly diagnosed multiple myeloma (NDMM) received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1 day 1, 56 mg/m² on cycle 1 days 8 and 15, and then 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- NDMM Dose-expansion: Carfilzomib 70 mg/m² (Experimental): Participants with NDMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone
- NDMM Dose-expansion: Carfilzomib 56 mg/m² (Experimental): Participants with NDMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 56 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Administered once weekly by 30-minute intravenous (IV) infusion on days 1, 8, and 15 of each 28-day cycle.
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
Drug: Lenalidomide — Administered orally once daily on days 1-21 of each 28-day cycle.
  Other Names: Revlimid®
Drug: Dexamethasone — Administered by mouth or IV at 40 mg on days 1, 8, and 15 of each 28-day cycle and on day 22 of cycles 1 to 8.

SUMMARY:
The purpose of the study is to assess the safety, tolerability and activity of a once-weekly regimen of carfilzomib in combination with lenalidomide and dexamethasone for the treatment of multiple myeloma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Newly diagnosed or relapsed multiple myeloma
2. Measureable disease by serum M protein, or urine M protein, or serum free light chain (SFLC) and an abnormal serum kappa lambda ratio (for subjects without detectable serum or urine M-protein), or serum quantitative immunoglobulin A (glgA) (for immunoglobulin (Ig) A subjects whose disease can only be reliable measured by qlgA).
3. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 to 2
4. Left ventricular ejection fraction (LVEF) ≥ 40%

Key Exclusion Criteria:

1. Waldenström macroglobulinemia
2. For newly diagnosed multiple myeloma: multiple myeloma of IgM subtype
3. For relapsed disease:

   1. If treated with a lenalidomide and dexamethasone combination, progression during the first 3 months after initiating treatment.
   2. Any progression during treatment if the lenalidomide and dexamethasone regimen was the most recent line of therapy.
   3. Any prior treatment with carfilzomib
4. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
5. Plasma cell leukemia (> 2.0 × 10^9/L circulating plasma cells by standard differential)
6. Myelodysplastic syndrome
7. Amyloidosis
8. Prior treatment with carfilzomib or oprozomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2019-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Kimball, MD, Study Director — Amgen
Locations (56):
- United States (56):
  - Research Site, Bakersfield, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Research Site, Burbank, California
  - Providence Saint Joseph Medical Center, Burbank, California
  - Research Site, Fountain Valley, California
  - Compassionate Care Research Group, Inc., Fountain Valley, California
  - Research Site, Los Angeles, California
  - Los Angeles Hematology / Oncology Medical Group, Los Angeles, California
  - Research Site, Whittier, California
  - Research Site, Aurora, Colorado
  - University of Colorado, Aurora, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Lombardi Cancer Center, Pediatric Hematology Oncology, Washington D.C., District of Columbia
  - Research Site, Fort Myers, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Research Site, Tampa, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Research Site, Boston, Massachusetts
  - Dana Farber Partners Cancer Care, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Research Site, New York, New York
  - Clinical Research Alliance, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Morton Coleman, MD, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Research Site, Stony Brook, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Research Site, Durham, North Carolina
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - Research Site, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Cincinnati, Ohio
  - Research Site, Bend, Oregon
  - Bend Memorial Clinic, Bend, Oregon
  - Research Site, Charleston, South Carolina
  - Medical University of South Carolina, Hollings Cancer Center, Charleston, South Carolina
  - Research Site, Greenville, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Saint Francis Hospital Cancer Center, Greenville, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Research Site, Germantown, Tennessee
  - The West Clinic, PC, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Tennessee Oncology, PLLC / The Sarah Cannon Research lnstitute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Research Site, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Aurora Health Care, Aurora Cancer Care, Milwaukee, Wisconsin
  - Research Site, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biran N, Siegel D, Berdeja JG, Raje N, Cornell RF, Alsina M, Kovacsovics T, Fang B, Kimball AS, Landgren O. Weekly carfilzomib, lenalidomide, and dexamethasone in relapsed or refractory multiple myeloma: A phase 1b study. Am J Hematol. 2019 Jul;94(7):794-802. doi: 10.1002/ajh.25498. Epub 2019 May 13. PMID 31021005
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 21 centers in the United States. The study had 2 parts: dose-evaluation and dose-expansion.
Pre-assignment Details: A Cohort Safety Review Committee (CSRC) reviewed all safety data and made recommendations regarding ongoing enrollment and opening of subsequent cohorts during the dose-evaluation component. The CSRC also selected the dose regimens evaluated in the dose-expansion component.
Period: Overall Study
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Started | 10 | 12 | 34 | 9 | 9 | 33
Completed | 2 | 3 | 2 | 0 | 1 | 1
Not Completed | 8 | 9 | 32 | 9 | 8 | 32
Not completed — Sponsor Decision | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 2 | 1 | 3 | 9
Not completed — Death | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Specified Criteria | 5 | 7 | 27 | 7 | 5 | 21

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m² | Total
Number analyzed (Participants) | 10 | 12 | 34 | 9 | 9 | 33 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.3) | 66.4 (8.1) | 61.9 (11.2) | 59.0 (14.0) | 61.8 (6.5) | 60.4 (10.7) | 61.7 (10.6)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 4 | 5 | 20 | 6 | 6 | 23 | 64
  65 to 74 years | 5 | 6 | 10 | 3 | 3 | 9 | 36
  ≥ 75 years | 1 | 1 | 4 | 0 | 0 | 1 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 15 | 3 | 3 | 16 | 45
  Male | 7 | 7 | 19 | 6 | 6 | 17 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 3 | 0 | 2 | 1 | 7
  Not Hispanic or Latino | 10 | 10 | 30 | 9 | 7 | 30 | 96
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 1 | 0 | 0 | 1 | 4
  Black or African American | 1 | 4 | 4 | 2 | 1 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 1
  White | 8 | 7 | 24 | 7 | 7 | 28 | 81
  Other | 0 | 0 | 4 | 0 | 1 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Safety and tolerability were evaluated according to the type, incidence, and severity of adverse events.
  An AE is defined as any untoward medical occurrence in a clinical trial subject. The event does not necessarily have a causal relationship with study treatment.
  A serious adverse event is defined as an AE that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening
  * requires in-patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
  The severity of each AE was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.03 where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening, and Grade 5 = Death.
Time Frame: From the first dose of any study drug up to 30 days after the last dose of any study drug; median (range) duration of treatment with carfilzomib was 32 (1.1, 76.7) weeks in RRMM participants and 26 (1.0, 94.4) weeks in NDMM participants.
Population: All participants who received at least 1 dose of study drug (safety analysis set).
Measure: Count of Participants; unit: Participants
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 9 | 9 | 33
Participants
  Any adverse event (AE) | 10 | 12 | 34 | 9 | 9 | 33
  AE Grade ≥ 3 | 7 | 9 | 23 | 5 | 6 | 21
  Serious adverse events | 4 | 5 | 10 | 3 | 3 | 11
  AEs leading to discontinuation of carfilzomib | 1 | 2 | 5 | 0 | 2 | 1
  AEs leading to discontinuation of lenalidomide | 1 | 2 | 5 | 0 | 2 | 2
  AEs leading to discontinuation of dexamethasone | 1 | 2 | 5 | 0 | 2 | 2
  Fatal adverse events | 0 | 0 | 2 | 0 | 0 | 0
  Treatment-related adverse events (TRAE) | 9 | 11 | 30 | 9 | 9 | 32
  Treatment-related AEs Grade ≥ 3 | 6 | 8 | 18 | 5 | 5 | 18
  Treatment-related serious adverse events | 1 | 2 | 6 | 1 | 3 | 8
  TRAEs leading to discontinuation of carfilzomib | 1 | 1 | 5 | 0 | 2 | 1
  TRAEs leading to discontinuation of lenalidomide | 1 | 1 | 5 | 0 | 2 | 2
  TRAEs leading to discontinuation of dexamethasone | 1 | 1 | 5 | 0 | 2 | 2
  Treatment-related fatal adverse events | 0 | 0 | 2 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Hemoglobin Levels
Time Frame: Baseline and Cycle 1, days 8 and 15 and Cycle 2 days 1, 8, and 15
Population: Participants in the safety analysis set with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 33
g/L
  Baseline | 116.90 (14.58) | 120.67 (13.51) | 123.24 (16.57) | 111.50 (18.04) | 120.00 (20.96) | 113.21 (16.66)
  Change from Baseline to Cycle 1 Day 8: number analyzed (Participants) | 10 | 12 | 33 | 8 | 9 | 33
  Change from Baseline to Cycle 1 Day 8 | -1.50 (7.52) | -3.33 (6.39) | -0.91 (5.46) | -1.25 (8.17) | -5.56 (6.11) | -1.82 (7.21)
  Change from Baseline to Cycle 1 Day 15: number analyzed (Participants) | 10 | 12 | 31 | 8 | 8 | 33
  Change from Baseline to Cycle 1 Day 15 | -6.90 (8.61) | -9.50 (6.29) | -5.10 (7.88) | -1.75 (12.70) | -6.50 (10.20) | -5.64 (9.10)
  Change from Baseline to Cycle 2 Day 1: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 1 | -5.70 (9.78) | -9.25 (8.67) | -7.38 (7.76) | -3.75 (12.65) | -3.29 (9.60) | 2.19 (10.59)
  Change from Baseline to Cycle 2 Day 8: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 8 | -6.00 (11.91) | -8.17 (9.00) | -5.59 (8.35) | -0.13 (14.64) | -2.86 (8.49) | 4.19 (12.41)
  Change from Baseline to Cycle 2 Day 15: number analyzed (Participants) | 10 | 12 | 31 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 15 | -8.50 (12.47) | -11.33 (8.04) | -8.45 (10.08) | 0.00 (14.05) | -5.14 (13.58) | 2.97 (13.04)

3. Primary Outcome: Change From Baseline in Platelet Count
Time Frame: Baseline and Cycle 1, days 8 and 15 and Cycle 2 days 1, 8, and 15
Population: Participants in the safety analysis set with available data at Baseline and each time point.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 33
10^9 cells/L
  Baseline | 151.60 (54.40) | 202.50 (67.13) | 172.38 (33.70) | 214.00 (79.22) | 242.89 (99.24) | 233.03 (67.76)
  Change from Baseline to Cycle 1 Day 8: number analyzed (Participants) | 10 | 12 | 33 | 8 | 9 | 33
  Change from Baseline to Cycle 1 Day 8 | -12.90 (29.88) | -49.50 (58.90) | -17.36 (21.75) | 2.38 (63.66) | -51.11 (42.10) | -21.42 (36.40)
  Change from Baseline to Cycle 1 Day 15: number analyzed (Participants) | 10 | 12 | 31 | 8 | 8 | 33
  Change from Baseline to Cycle 1 Day 15 | -58.60 (32.76) | -66.83 (87.14) | -66.39 (38.30) | -23.25 (116.67) | -101.88 (84.66) | -53.39 (43.60)
  Change from Baseline to Cycle 2 Day 1: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 1 | 55.00 (38.61) | 68.67 (84.62) | 44.84 (52.82) | 141.75 (92.68) | 152.00 (244.50) | 111.06 (84.26)
  Change from Baseline to Cycle 2 Day 8: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 8 | -44.10 (38.14) | -74.75 (86.91) | -71.06 (37.93) | -28.00 (111.10) | -106.29 (130.18) | -52.78 (60.70)
  Change from Baseline to Cycle 2 Day 15: number analyzed (Participants) | 10 | 12 | 31 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 15 | -44.40 (21.48) | -63.25 (72.53) | -60.13 (43.37) | -21.25 (82.11) | -76.14 (116.02) | -44.19 (64.73)

4. Primary Outcome: Change From Baseline in Neutrophil Count
Time Frame: Baseline and Cycle 1, days 8 and 15 and Cycle 2 days 1, 8, and 15
Population: Participants in the safety analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 33
10^9 cells/L
  Baseline | 2.53 (1.01) | 3.40 (1.54) | 2.72 (0.94) | 3.04 (0.73) | 3.24 (2.24) | 3.26 (1.46)
  Change from Baseline to Cycle 1 Day 8: number analyzed (Participants) | 10 | 12 | 33 | 8 | 9 | 33
  Change from Baseline to Cycle 1 Day 8 | 0.02 (0.82) | 0.03 (1.87) | 0.97 (1.19) | 0.59 (1.20) | -0.19 (1.25) | 0.37 (1.29)
  Change from Baseline to Cycle 1 Day 15: number analyzed (Participants) | 10 | 12 | 28 | 8 | 8 | 33
  Change from Baseline to Cycle 1 Day 15 | 0.28 (1.14) | -0.09 (1.94) | 0.81 (1.09) | 1.08 (1.53) | 0.43 (1.83) | 0.09 (1.48)
  Change from Baseline to Cycle 2 Day 1: number analyzed (Participants) | 10 | 12 | 31 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 1 | 0.36 (1.99) | -0.33 (1.59) | 0.16 (1.15) | 0.02 (0.58) | 0.09 (2.46) | 0.18 (0.95)
  Change from Baseline to Cycle 2 Day 8: number analyzed (Participants) | 9 | 12 | 29 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 8 | 0.18 (0.68) | -0.67 (1.28) | 0.63 (1.08) | 0.57 (1.05) | 0.46 (2.49) | 0.41 (1.25)
  Change from Baseline to Cycle 2 Day 15: number analyzed (Participants) | 10 | 11 | 31 | 8 | 7 | 32
  Change from Baseline to Cycle 2 Day 15 | -0.30 (0.71) | -0.54 (1.69) | -0.06 (1.25) | 0.33 (0.53) | 0.56 (2.92) | 0.42 (2.00)

5. Primary Outcome: Change From Baseline in Bilirubin
Time Frame: Baseline and Cycle 2 day 1
Population: Participants in the safety analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 33
µmol/L
  Baseline: number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 32
  Baseline | 8.55 (3.78) | 9.98 (4.72) | 9.10 (4.76) | 10.26 (4.38) | 6.84 (4.01) | 7.16 (3.29)
  Change from Baseline to Cycle 2 Day 1: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 31
  Change from Baseline to Cycle 2 Day 1 | 0.86 (3.25) | 1.00 (3.68) | 1.34 (3.52) | 3.42 (5.56) | 0.49 (2.91) | 1.21 (3.10)

6. Primary Outcome: Change From Baseline in Creatinine
Time Frame: Baseline and Cycle 1, days 8 and 15 and Cycle 2 days 1, 8, and 15
Population: Participants in the safety analysis set with available data at each time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 33
µmol/L
  Baseline: number analyzed (Participants) | 10 | 12 | 34 | 8 | 9 | 32
  Baseline | 80.18 (18.57) | 82.88 (22.01) | 79.09 (17.61) | 75.80 (7.78) | 95.37 (41.17) | 80.60 (21.56)
  Change from Baseline to Cycle 1 Day 8: number analyzed (Participants) | 10 | 10 | 33 | 8 | 8 | 32
  Change from Baseline to Cycle 1 Day 8 | -2.65 (5.05) | -5.30 (10.29) | 2.09 (8.31) | -1.22 (8.25) | -8.51 (29.44) | -0.22 (12.89)
  Change from Baseline to Cycle 1 Day 15: number analyzed (Participants) | 9 | 10 | 31 | 8 | 8 | 32
  Change from Baseline to Cycle 1 Day 15 | -4.42 (7.92) | -4.60 (11.32) | -1.85 (12.69) | 3.65 (27.29) | 29.39 (130.24) | 0.42 (17.59)
  Change from Baseline to Cycle 2 Day 1: number analyzed (Participants) | 10 | 12 | 32 | 8 | 7 | 31
  Change from Baseline to Cycle 2 Day 1 | -3.80 (6.81) | -7.74 (11.98) | -1.44 (9.66) | -10.39 (10.05) | -17.17 (36.71) | -4.31 (9.84)
  Change from Baseline to Cycle 2 Day 8: number analyzed (Participants) | 10 | 11 | 32 | 8 | 7 | 31
  Change from Baseline to Cycle 2 Day 8 | -6.45 (4.97) | -11.09 (12.70) | 1.85 (10.95) | -12.27 (8.20) | -20.08 (37.86) | -4.32 (9.36)
  Change from Baseline to Cycle 2 Day 15: number analyzed (Participants) | 10 | 12 | 31 | 8 | 7 | 31
  Change from Baseline to Cycle 2 Day 15 | -6.28 (10.29) | -13.26 (9.05) | 4.88 (13.78) | -12.38 (6.90) | -21.85 (39.17) | -1.99 (18.08)

7. Secondary Outcome: Maximum Plasma Concentration of Carfilzomib on Day 8 of Cycle 1 by Dose Group
Time Frame: Day 8 of Cycle 1 at predose, 15 minutes after the start of infusion, at the end of infusion, and 15 and 60 minutes after the end of infusion
Population: Participants who received at least 1 dose of study drug who had sufficient carfilzomib exposure and plasma concentration versus time data for the estimation of pharmacokinetic parameters by a non-compartmental analysis on day 8 of cycle 1.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Carfilzomib 56 mg/m²: Participants who received carfilzomib 56 mg/m² on Cycle 1 day 8.
- Carfilzomib 70 mg/m²: Participants who received carfilzomib 70 mg/m² on Cycle 1 day 8.
Arm/Group | Carfilzomib 56 mg/m² | Carfilzomib 70 mg/m²
Number analyzed (Participants) | 46 | 40
ng/mL | 11700 (67300) | 12400 (45000)

8. Secondary Outcome: Time to Maximum Plasma Concentration of Carfilzomib on Day 8 of Cycle 1 by Dose Group
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Carfilzomib 56 mg/m² | Carfilzomib 70 mg/m²
Number analyzed (Participants) | 46 | 40
hours | 0.28 [0.17 to 24] | 0.27 [0.17 to 0.68]

9. Secondary Outcome: Area Under the Curve From Time Zero to Time of Last Quantifiable Concentration of Carfilzomib on Day 8 of Cycle 1 by Dose Group
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Carfilzomib 56 mg/m² | Carfilzomib 70 mg/m²
Number analyzed (Participants) | 46 | 40
hr*ng/mL | 4150 (17500) | 9130 (32800)

10. Secondary Outcome: Overall Response Rate (ORR)
Description: Response was determined by the investigator based on the International Myeloma Working Group Uniform Response Criteria (IMWG URC). ORR was defined as the percentage of participants who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). Responses must have been confirmed in 2 consecutive assessments at any time prior to initiation of any new therapy.
  Disease assessments included serum protein electrophoresis (SPEP) with immunofixation, urine protein electrophoresis (UPEP; 24-hour assessment) with immunofixation, serum free light chain (SFLC), quantitative immunoglobulins, bone marrow aspirates to determine percent plasma cell involvement, and skeletal imaging for plasmacytoma evaluation.
Time Frame: Response assessments were performed on day 1 of each treatment cycle from cycle 2 and then every 8 weeks during follow-up until disease progression. Median time on follow-up was 10.6 months in RRMM participants and 6.9 months in NDMM participants.
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- RRMM: Combined Carfilzomib 70 mg/m²: Participants with RRMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, and 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
- NDMM: Combined Carfilzomib 70 mg/m²: Participants with NDMM received treatment with carfilzomib, lenalidomide, and dexamethasone (KRd) for up to eighteen 28-day cycles, or until disease progression, patient withdrawal, stem cell transplant, or death.
  Participants received carfilzomib on days 1, 8, and 15 of each cycle. The dose was 20 mg/m² on cycle 1, day 1, 56 or 70 mg/m² on cycle 1 days 8 and 15, and 70 mg/m² thereafter. Participants also received lenalidomide 25 mg once daily on days 1-21 and dexamethasone 40 mg (oral or IV) on days 1, 8, and 15 of each cycle, and on day 22 of cycles 1 to 8.
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | RRMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 46 | 9 | 9 | 18 | 33
percentage of participants | 90.0 [55.5 to 99.7] | 91.7 [61.5 to 99.8] | 88.2 [72.5 to 96.7] | 89.1 [76.4 to 96.4] | 88.9 [51.8 to 99.7] | 77.8 [40.0 to 97.2] | 83.3 [58.6 to 96.4] | 97.0 [84.2 to 99.9]

11. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete Response Rate (CRR) is defined as the percentage of participants who achieved a best overall response of either stringent complete response (sCR) or complete response (CR) in accordance with International Myeloma Working Group-Uniform Response Criteria (IMWG-URC).
  sCR: As for CR, and absence of clonal plasma cells in bone marrow (BM) CR: Negative serum and urine immunofixation, disappearance of any soft tissue plasmacytomas, < 5% plasma cells in BM, and normal SFLC ratio in participants with measurable disease only by SFLC.
Time Frame: as for outcome 10
Population: Participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | RRMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 46 | 9 | 9 | 18 | 33
percentage of participants | 20.0 [2.5 to 55.6] | 16.7 [2.1 to 48.4] | 26.5 [12.9 to 44.4] | 23.9 [12.6 to 38.8] | 22.2 [2.8 to 60.0] | 11.1 [0.3 to 48.2] | 16.7 [3.6 to 41.4] | 33.3 [18.0 to 51.8]

12. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first day of study treatment to the earlier of disease progression or death due to any cause.
  Disease progression was determined by the investigator according to IMWG-URC. Progressive Disease (PD): Increase of 25% from lowest value in serum M-component (absolute increase ≥ 0.5 g/dL), urine M-component (absolute increase ≥ 200 mg per 24 hours) and/or the difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL) in patients without measurable serum and urine M-protein levels, and/or any new or increase in size of bone lesions or soft tissue plasmacytomas, or development of hypercalcemia.
  PFS was analyzed using Kaplan-Meier methods. Participants who were alive with no documented PD, started new anticancer therapy before documentation of PD or death, had death or PD immediately after > 1 consecutively missed assessment visit, were lost to follow-up or withdrew consent were censored at the date of last disease assessment.
Time Frame: From first dose of study drug until the end of follow-up; Median time on follow-up was 10.6 months in RRMM participants and 6.9 months in NDMM participants.
Population: Participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | RRMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 10 | 12 | 34 | 46 | 9 | 9 | 18 | 33
months | NA [14.8 to NA] — Could not be estimated due to the low number of events | NA [5.6 to NA] — Could not be estimated due to the low number of events | NA [21.1 to NA] — Could not be estimated due to the low number of events | NA [21.1 to NA] — Could not be estimated due to the low number of events | NA [4.7 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

13. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response (DOR) was calculated for participants who achieved a confirmed PR or better based on Investigator assessment and according to the IMWG URC. Duration of overall response is defined as the time from first documentation of response to disease progression or death due to any cause. DOR was analyzed using Kaplan-Meier methods. Participants who were alive with no documented PD, started new anticancer therapy before documentation of PD or death, had death or PD immediately after > 1 consecutively missed disease assessment visit, were lost to follow-up, or withdrew consent were censored at the date of last disease assessment.
Time Frame: as for outcome 12
Population: Participants who received at least 1 dose of study drug with an overall response of PR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | RRMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM: Combined Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
Number analyzed (Participants) | 9 | 11 | 30 | 41 | 8 | 7 | 15 | 32
months | NA [NA to NA] — Could not be estimated due to the low number of events | NA [11.6 to NA] — Could not be estimated due to the low number of events | NA [20.2 to NA] — Could not be estimated due to the low number of events | NA [20.2 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

ADVERSE EVENTS:
Time Frame: All-cause Mortality is reported from the enrollment date up to the end of study; maximum time on study was 30.6 months. Treatment-emergent adverse events are reported from the first dose of any study drug up to 30 days after the last dose of any study drug; median (range) duration of treatment with carfilzomib was 32 (1.1, 76.7) weeks in RRMM participants and 26 (1.0, 94.4) weeks in NDMM participants.
Arm/Group | RRMM Dose-evaluation: Carfilzomib 56 mg/m² | RRMM Dose-evaluation: Carfilzomib 70 mg/m² | RRMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² | NDMM Dose-expansion: Carfilzomib 70 mg/m² | NDMM Dose-expansion: Carfilzomib 56 mg/m²
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 2/34 | 0/9 | 0/9 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/10 | 5/12 | 10/34 | 3/9 | 3/9 | 11/33
Other Adverse Events (participants affected / at risk) | 10/10 | 12/12 | 33/34 | 9/9 | 9/9 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RRMM Dose-evaluation: Carfilzomib 56 mg/m² (N=10) | RRMM Dose-evaluation: Carfilzomib 70 mg/m² (N=12) | RRMM Dose-expansion: Carfilzomib 70 mg/m² (N=34) | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² (N=9) | NDMM Dose-expansion: Carfilzomib 70 mg/m² (N=9) | NDMM Dose-expansion: Carfilzomib 56 mg/m² (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Vitello-intestinal duct remnant (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Strangulated hernia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RRMM Dose-evaluation: Carfilzomib 56 mg/m² (N=10) | RRMM Dose-evaluation: Carfilzomib 70 mg/m² (N=12) | RRMM Dose-expansion: Carfilzomib 70 mg/m² (N=34) | NDMM Dose-evaluation: Carfilzomib 56/70 mg/m² (N=9) | NDMM Dose-expansion: Carfilzomib 70 mg/m² (N=9) | NDMM Dose-expansion: Carfilzomib 56 mg/m² (N=33)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 9 | 1 | 2 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 4 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 4 | 6 | 0 | 1 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 3 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 2 | 2 | 0 | 1 | 1
Eye disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Halo vision (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 2 | 4 | 1 | 1 | 3
Visual impairment (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2 | 1 | 0 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 2
Chapped lips (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 7 | 7 | 5 | 2 | 10
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 18 | 7 | 6 | 16
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 3 | 0 | 1 | 8
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Food poisoning (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 2 | 12 | 2 | 4 | 17
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Palatal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 6 | 1 | 1 | 6
Administration site oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 2 | 0 | 1 | 0 | 3
Chest discomfort (General disorders) | 1 | 1 | 3 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 4 | 1 | 0 | 2
Chills (General disorders) | 1 | 1 | 2 | 0 | 1 | 2
Cyst (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Energy increased (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 4 | 21 | 3 | 4 | 13
Gait disturbance (General disorders) | 0 | 1 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 3 | 1 | 0 | 1
Injection site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 2 | 1
Malaise (General disorders) | 1 | 1 | 1 | 0 | 0 | 2
Mucosal inflammation (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 4 | 4 | 2 | 11
Pain (General disorders) | 2 | 1 | 1 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 2 | 0 | 0 | 3
Pyrexia (General disorders) | 5 | 2 | 5 | 1 | 3 | 6
Swelling (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Swelling face (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Thirst (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Immune system disorder (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Implant site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 1 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 6
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 4 | 2 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 7 | 14 | 3 | 1 | 15
Urinary tract infection (Infections and infestations) | 0 | 1 | 3 | 1 | 1 | 3
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 1 | 4 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 3 | 1 | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 3 | 0 | 0 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 5
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 2 | 5 | 1 | 0 | 3
Blood creatinine increased (Investigations) | 1 | 1 | 4 | 1 | 0 | 1
Blood uric acid decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 2 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Globulins increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 2 | 1 | 0 | 3
Neutrophil count decreased (Investigations) | 2 | 0 | 4 | 2 | 0 | 3
Platelet count decreased (Investigations) | 1 | 3 | 11 | 2 | 0 | 3
Weight decreased (Investigations) | 0 | 1 | 2 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 5 | 1 | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 4 | 2 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 3 | 0 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 5 | 0 | 0 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3 | 1 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 8 | 4 | 0 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0 | 5
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 0 | 1 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 8 | 4 | 2 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 6 | 10 | 2 | 3 | 8
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 9 | 2 | 2 | 12
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 4 | 1 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1 | 1 | 2
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 5
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 1 | 2 | 6
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 7 | 3 | 1 | 12
Dysgeusia (Nervous system disorders) | 0 | 3 | 0 | 0 | 2 | 7
Headache (Nervous system disorders) | 1 | 3 | 8 | 3 | 5 | 13
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 3 | 2 | 2 | 4
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 3 | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 3 | 1 | 1 | 5
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Taste disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1
Tremor (Nervous system disorders) | 2 | 2 | 2 | 0 | 0 | 5
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 4
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 4
Depression (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3 | 7 | 2 | 0 | 17
Irritability (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 4
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 4
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 2 | 0 | 1 | 3
Urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 11 | 4 | 2 | 12
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 9 | 2 | 1 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 0 | 2 | 1
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 1 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 6 | 0 | 1 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 2 | 1 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 3
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 5 | 1 | 2 | 11
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 5 | 4 | 4 | 8
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 2 | 0 | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 4 | 7 | 1 | 2 | 1
Hypotension (Vascular disorders) | 2 | 0 | 2 | 1 | 0 | 2
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 2
Vascular pain (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vein discolouration (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT02335983/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02335983/SAP_001.pdf